CLINICAL TRIAL: NCT00173771
Title: Development of a Comprehensive ADL Scale for Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9361701233; NSC-94-2314-B-002-076
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-08

CONDITIONS: Cerebrovascular Accidents
Keywords: stroke; activities of daily living; psychometrics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
our research team will develop a new CADL scale for stroke patients over the next three years.

In the first year, we had established a CADL item bank of 50 items. The investigators will administer the 50 items on 300 patients with stroke living in the community. Then we will select 10 to 15 items from the item bank for the CADL scale based on the International Classification of Functioning, Disability and Health (ICF), the opinions of an expert panel, and Rasch analysis. It is anticipated that the CADL scale will have unidimensionality, an interval level of measurement, soundly psychometric characteristics, a reduced number of items, and ease of administration.

In the second and third years, we will compare the psychometric properties of the CADL scale and the combined BI and FAI scale. The psychometric properties investigated will include reliability (e.g. inter-rater reliability, intra-rater reliability, and internal consistency), validity (e.g. concurrent validity, convergent validity, predictive validity and discriminant validity), and responsiveness. A total of 150 patients will be recruited. Both the CADL scale and the combined BI and FAI scale will be used on patients from the initial stage (within one month) to six months after hospital discharge. The results will be useful for researchers and clinicians to determine whether the CADL scale is better than the combined BI and FAI scale in stroke patients.

DETAILED DESCRIPTION:
our research team will develop a new CADL scale for stroke patients over the next three years.

In the first year (an ongoing project: NSC 93-2314-B-002-284), we had established a CADL item bank of 50 items. The investigators will administer the 50 items on 300 patients with stroke living in the community. Then we will select 10 to 15 items from the item bank for the CADL scale based on the International Classification of Functioning, Disability and Health (ICF), the opinions of an expert panel, and Rasch analysis. It is anticipated that the CADL scale will have unidimensionality, an interval level of measurement, soundly psychometric characteristics, a reduced number of items, and ease of administration.

In the second and third years, we will compare the psychometric properties of the CADL scale and the combined BI and FAI scale. The psychometric properties investigated will include reliability (e.g. inter-rater reliability, intra-rater reliability, and internal consistency), validity (e.g. concurrent validity, convergent validity, predictive validity and discriminant validity), and responsiveness. A total of 150 patients will be recruited. Both the CADL scale and the combined BI and FAI scale will be used on patients from the initial stage (within one month) to six months after hospital discharge. The results will be useful for researchers and clinicians to determine whether the CADL scale is better than the combined BI and FAI scale in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

diagnosis of stroke

Exclusion Criteria:

with other major diseases (e.g., cancer)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2004-08; Study Completion 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: I-Ping Hsueh, MA, Principal Investigator — School of Occupational Therapy, College of Medicine, National Taiwan University
Locations (1):
- School of Occupational Therapy, College of Medicine, National Taiwan University, Dawan, Taiwan